CLINICAL TRIAL: NCT03247907
Title: Humidification Needs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was terminated by investigators due to equipment difficulties
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CIA-191
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Condition A: CPAP with No Humidification (Active Comparator): CPAP with No Humidification with no mouth leak
  Interventions: Device: Condition A: CPAP with No Humidification
- Condition B: CPAP with No Humidification (Active Comparator): CPAP with No Humidification with mouth leak
  Interventions: Device: Condition B: CPAP with No Humidification
- Condition C: CPAP with Cold Passover humidifier (Active Comparator): CPAP with Cold Passover humidifier with mouth leak
  Interventions: Device: Condition C: CPAP with Cold Passover
- Condition D: CPAP with Modified Humidifier (Active Comparator): CPAP with Modified Humidifier with mouth leak
  Interventions: Device: Condition D: CPAP with Modified humidifier
- Condition E: CPAP with Ambient Tracking (Active Comparator): CPAP with Ambient Tracking with mouth leak
  Interventions: Device: Condition E: CPAP with Ambient Tracking
- Condition F: CPAP with Heated Humidification (Active Comparator): CPAP with Heated Humidification at default setting with mouth leak
  Interventions: Device: Condition F: CPAP with Heated Humidification
- Condition G: CPAP with Heated Humidification (Active Comparator): CPAP with Heated Humidification at max setting with mouth leak
  Interventions: Device: Condition G: CPAP with Heated Humidification
- Condition H: CPAP with New level humidification (Active Comparator): CPAP with New level humidification with mouth leak
  Interventions: Device: Condition H: CPAP with New level humidification

INTERVENTIONS:
Device: Condition A: CPAP with No Humidification — CPAP with No Humidification with no mouth leak
  Arms: Condition A: CPAP with No Humidification
Device: Condition B: CPAP with No Humidification — CPAP with No Humidification with mouth leak
  Arms: Condition B: CPAP with No Humidification
Device: Condition C: CPAP with Cold Passover — CPAP with Cold Passover with mouth leak
  Arms: Condition C: CPAP with Cold Passover humidifier
Device: Condition D: CPAP with Modified humidifier — CPAP with Modified humidifier with mouth leak
  Arms: Condition D: CPAP with Modified Humidifier
Device: Condition E: CPAP with Ambient Tracking — CPAP with Ambient Tracking with mouth leak
  Arms: Condition E: CPAP with Ambient Tracking
Device: Condition F: CPAP with Heated Humidification — CPAP with Heated Humidification at default setting with mouth leak
  Arms: Condition F: CPAP with Heated Humidification
Device: Condition G: CPAP with Heated Humidification — CPAP with Heated Humidification at max setting with mouth leak
  Arms: Condition G: CPAP with Heated Humidification
Device: Condition H: CPAP with New level humidification — CPAP with New level humidification with mouth leak
  Arms: Condition H: CPAP with New level humidification

SUMMARY:
A study undertaken to investigate mouth leak for airway discomfort/dryness while using CPAP. This study will also measure how much humidification is required to treat subsequent upper airway discomfort/dryness from mouth leak by utilizing different levels and types of humidification.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over

Exclusion Criteria:

* Inability to give consent
* Currently pregnant or think they may be pregnant
* Current nasal symptoms or chronic nasal disease
* Contraindicated for PAP therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Nasal Resistance | 8 Days
  Will be measured by rhinomanometer or acoustic rhinometry
Evaluation of Nasal Dryness and Discomfort | 8 Days
  Reported by participants using the Xero Questionnaire

SECONDARY OUTCOMES:
Preference of Testing Condition | 8 Days
  Measured by custom preference questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher and Paykel Healthcare, East Tamaki, Auckland, New Zealand